CLINICAL TRIAL: NCT02175498
Title: A Clinical Study to Assess the Effectiveness of Homeopathic Treatment in Female Infertility
Brief Title: Effectiveness of Homeopathic Treatment in Female Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Collaborators: Father Muller Medical College (Other)
Responsible Party: Principal Investigator, Dr Anita Fernandes, Principal Investigator, Fr Muller Homoeopathic Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APB123
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Female Infertility
Keywords: Homoeopathy Similimum female infertility
MeSH Terms: conditions — Infertility, Female | interventions — Homeopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Homoeopathic medicines (Experimental): 4 pills once a week of the indicated similium for a period of one year
  Interventions: Drug: Homoeopathic medicines

INTERVENTIONS:
Drug: Homoeopathic medicines — 4 pills once a week of the indicated Similimum
  Other Names: indicated Homoeopathic similimum

SUMMARY:
The purpose of this study is to assess the effectiveness of Homoeopathic treatment in female infertility.

DETAILED DESCRIPTION:
Objectives:

• To assess the rate of conception, in female infertility, after individualized homoeopathic treatment.

Need for the study:

* To confirm that homeopathy is best alternative for resource limited community to receive effective treatment with minimum possible expenditure.
* To bring out a repertoire of effective Homoeopathic medicines in the treatment of infertility.
* To establish a centre for focussed treatment of infertility at Father Muller Homeopathic Medical College and Hospital.

Many cases visiting Homoeopathic OPD have improved under the treatment. In general, there is a deficit of well-designed, randomized, controlled trials to evaluate the efficacy and safety of complementary and alternative medicine for these indications, which makes it difficult to provide evidence-based recommendations.

Globally there is a need for this study to avoid the side-effects of antibiotics and hormonal tablets thus improving the quality of life. In a third world country like India where infertile females cannot afford surgery; Homoeopathic medicines are simple, safe and cost effective. Homoeopathy can treat the underlying cause of female infertility in these cases and thereby prevent the hazards of surgery. In India the female race is always targeted and blamed for being infertile. This not only has an impact on the health of the woman but also affects her social status. The psychological and mental agony suffered by these infertile women and the fear that their husbands' may go in for a second marriage in turn causes great stress and anxiety. Hence the efficacy of Homoeopathic medicines on infertile females needs to be explored.

Methodology:

Approach: This is a prospective study with purposive sampling. Design: Total number of beneficiaries is 40, including 20 PCOS cases, 10 cases of Endometriosis, and 10 cases of Chronic Pelvic Inflammatory diseases. The numbers of these cases are based on the availability and frequency of their visits to our OPD.

Data collection instruments: case books of the OPD Setting: OPD of Homeopathic Medical College, Derlakatte, Kankanady and Thumbe Population: women visiting the OPD for infertility treatment Sample: women diagnosed for any of the three causes of infertility Sampling technique: purposive sampling Feasibility: the study is feasible in terms of availability of patients at our OPD settings Duration of study: total of 3 years. All 40 cases are expected to be registered in a span of 6 months to 1 year. Registration will be followed by treatment of 18 months, 6 months for analysis and reporting by the end of 3 years.

Statistical analysis: Data from the sample is collected and subjected to chi square test, and frequencies will be calculated.

Null Hypothesis: No significant difference in cases of female infertility before and after treatment.

Alternate Hypothesis: Significant difference in cases of female infertility before and after treatment.

Procedure:

Forty infertile women will undergo investigations like Ultrasonography of pelvis, diagnostic laparoscopy when needed and urine pregnancy test once in six months. The cases will be diagnosed by the principal investigators and co-investigators. Semen analysis in male partners will be done as a routine to rule out cases of male infertility. The infertile women will be administered appropriate Homoeopathic Simillimum by the principal investigator for 18 months. The follow-up visits of these patients will be once in two weeks. Effectiveness of Homoeopathic treatment and rate of conception in infertile females will be assessed after administering the Simillimum. The investigations will be repeated after treatment and cases will be reviewed and examined by the co-investigators.

The treatment given is individually chosen homoeopathic medicine based on the psychophysical symptom syndrome each experienced. The drugs are procured from Fr Muller HPD which complies with the standards of Homoeopathic Pharmacopoeia. The investigations will be repeated after treatment.

The Homoeopathic treatment includes a detailed interview in which the patient is queried about her unique symptoms. The well indicated constitutional remedy will be given on the basis of symptoms' similarity, that is, symptoms that were in emotional and mental realm and those that affected her entire body. The symptoms will be ordered by intensity and prominence. A single dose of Homoeopathic Similimum will be given to each of these patients and repeated as and when needed and whenever required the potency will be increased. If there is any miasmatic block, anti-miasmatic treatment will be given. Acute remedy will be given when needed. All cases of infertility are told to abstain from caffeine and Allopathic treatment. Hormonal treatment is to be withdrawn. The investigations will be repeated after treatment after six months, twelve months and eighteen months whenever required to assess the improvement of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Only female causes
  * Age group of 18-40 years
  * Cases of PCOS, Endometriosis and Chronic PID
  * Primary and secondary infertility

Exclusion Criteria:

* Age group below 18 years and beyond 40 years
* All other causes such as unknown infertility, congenital defects
* Women whose husband's semen analysis is abnormal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Improved fertility rate | 3 years
  Investigative parameters becoming normal

SECONDARY OUTCOMES:
Positive pregnancy test | 3 years
  Earlie Icon

OTHER OUTCOMES:
Conception | 3 years
  Live intra-uterine foetus

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anita Fernandes, MD(HOM), Principal Investigator — Fr Muller Homoeopathic Medical College
Locations (1):
- Fr Muller Homoeopathic Medical College, Mangalore, Karnataka, India